CLINICAL TRIAL: NCT05430893
Title: Intra-muscular Botulinum Toxin A in Chronic Athletic Pubalgia: a Retrospective Observational Study
Brief Title: Intra-muscular Botulinum Toxin A in Chronic Athletic Pubalgia
Acronym: PUBATOX
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220617
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Athletic Pubalgia
Keywords: Chronic athletic pubalgia; Botulinum toxin; Groin pain; Adductor enthesopathy
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Athletic pubalgia: Patients with chronic athletic pubalgia for whom medical and/or surgical treatments have failed and who were treated with an intra-muscular injection of botulinum toxin A injection under ultrasound guidance
  Interventions: Other: Botulinum Toxin A

INTERVENTIONS:
Other: Botulinum Toxin A — 100 UI IM in the adductor longus

SUMMARY:
Chronic athletic pubalgia is a frequent sport condition in which the effectiveness of medical treatment has not been proven. Intra-muscular injection of botulinum toxin A may have positive effects on pain in some chronic tendinitis.

The investigators hypothesized that similar analgesic effect of intra-muscular botulinum toxin A may be observed in individuals with chronic AP. In the present study, the investigators aimed to describe the short-term evolution of pain and of activity limitations and quality of life, after an injection of the adductor longus with botulinum toxin A, in individuals with chronic AP, for whom medical and/or surgical treatments have failed.

DETAILED DESCRIPTION:
The investigators included consecutive individuals with chronic athletic pubalgia for whom medical and/or surgical treatments have failed and who were treated with an intra-muscular injection of botulinum toxin A under ultrasound guidance. Participants were assessed 50 days after injection for pain using a numerical rating scale (NRS) (0, no pain, and 100, maximal pain) and for activity limitations and quality of life using the Copenhagen Hip and Groin Outcome Score (HAGOS) (0, worse outcome, and 100, most favorable outcome). Participants were also asked to self-report adverse events.

ELIGIBILITY:
Inclusion Criteria:

* chronic AP
* symptom duration ≥ 3 months
* consistent clinical and magnetic resonance imaging findings according to the clinician
* failure of medical and/or surgical treatments with persistent pain and inability to return to play
* treatment with an intra-muscular injection of botulinum toxin A injection

Exclusion Criteria:

* age under 18 years
* ongoing pregnancy or breastfeeding
* treatments by anticoagulants
* muscular disorder (e.g. polymyositis, myopathy or other neuromuscular conditions)
* guardianship or curatorship
* individuals who had received botulinum toxin type A treatment for less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic athletic pubalgia for whom medical and/or surgical treatments have failed and who were treated with an intra-muscular injection of botulinum toxin A injection under ultrasound guidance
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale | 50 days
  Mean pain

SECONDARY OUTCOMES:
HAGOS score | 50 days
  Mean HAGOS total score

CONTACTS AND LOCATIONS:
Overall Officials: Romain GAROFOLI, Principal Investigator — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP); Marie-Martine Lefevre-Colau, MD, PhD, Study Director — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP)
Locations (1):
- Service de rééducation fonctionnelle, réadaptation de l'appareil locomoteur et Pathologies du Rachis - Cochin Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No